CLINICAL TRIAL: NCT01254942
Title: Mobilizing Evidence Into Action to Improve Outcomes of Vulnerable Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Maureen C. Ashe, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H09-01291
Record Dates: First submitted 2010-12-02; First posted 2010-12-07 (Estimated); Results first posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Hip Fractures; Femoral Fractures
Keywords: exercise; hip fractures; rehabilitation; aged; aged 80 and over
MeSH Terms: conditions — Hip Fractures; Femoral Fractures; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Usual care following hip fracture
  Interventions: Other: Usual Care
- Intervention (Experimental): Follow-up Fracture Clinic
  Interventions: Other: B4 Clinic

INTERVENTIONS:
Other: B4 Clinic — Fracture Follow-Up Clinic plus Exercise Program
  Arms: Intervention
Other: Usual Care
  Other Names: usual care pathways for after hip fracture
  Arms: Usual Care

SUMMARY:
This is a parallel Randomized Controlled Trial comparing two different delivery modes of post hip fracture management-a specialized Fracture Follow-up Clinic versus Usual Care alone. The Fracture Follow-up Clinic will focus on bone health and fall risk factors. The investigators will evaluate the effect of the clinic and exercise program on mobility and falls. The investigators primary hypothesis is that within the first year following a hip fracture, older adults who are assessed in the B4 Clinic and prescribed an exercise program will have significantly improved Short Physical Performance Battery (SPPB) scores compared with participants who receive usual care alone.

ELIGIBILITY:
Inclusion Criteria:

* 65 years +
* community-dwelling
* residents of Metro Vancouver
* recent history (within 12 months) of femoral fracture

Exclusion Criteria:

* unable to ambulate 10 meters prior to the femoral fracture were(with/without a walking aid)
* discharged to a residential care facility
* and/or diagnosed with any type of dementia (Alzheimer's, vascular etc.)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen C. Ashe, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia - VCHRI, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook WL, Khan KM, Bech MH, Brasher PM, Brown RA, Bryan S, Donaldson MG, Guy P, Hanson HM, Leia C, Macri EM, Sims-Gould J, McKay HA, Ashe MC. Post-discharge management following hip fracture--get you back to B4: a parallel group, randomized controlled trial study protocol. BMC Geriatr. 2011 Jun 9;11:30. doi: 10.1186/1471-2318-11-30. PMID 21651819
- [Result] Cook WL, Brasher PMA, Guy P, Bryan S, Donaldson MG, Sims-Gould J, McKay HA, Khan KM, Ashe MC. Comprehensive Geriatric Care to Improve Mobility after Hip Fracture: An RCT. Gerontology. 2020;66(6):542-548. doi: 10.1159/000510903. Epub 2020 Nov 11. PMID 33176306
- [Derived] Ashe MC, Grover S, Bryan S, Cook WL, Donaldson MG, Brasher PMA. Perceived Health Status and Capability after Hip Fracture: Secondary Outcomes from an Randomized Controlled Trial. Gerontology. 2024;70(3):235-240. doi: 10.1159/000536131. Epub 2024 Jan 5. PMID 38185111
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual care following hip fracture provided by the public health care system. this may include publicly funded home care services, rehab, and follow-up visits with doctors.
  Usual Care
- Intervention: Follow-up Fracture Clinic
  B4 Clinic: Fracture Follow-Up Clinic plus Exercise Program This is an interdisciplinary outpatient clinic within the public health care system. Participants were assessed by a geriatrician, physiotherapist, occupational therapist, and other health providers as needed. Management and sessions were determined by health providers and participants.
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 27 | 26
Completed | 25 | 24
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Usual care following hip fracture
  Usual Care
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 27 | 26 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  Canada | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Short Physical Performance Battery
Description: The primary outcome for this trial is the Short Physical Performance Battery (SPPB). The SPPB is composed of three separate tests that are timed and categorized depending on performance. The three domains evaluated in the SPPB are standing balance, gait speed, and sit to stand performance.
  The SPPB scores can range from 0-12, a higher score indicates better performance. The subscales are combined.
Time Frame: 12 months post-fracture
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 25 | 24
score on a scale | 8.24 (2.44) | 9.08 (3.03)

2. Secondary Outcome: Difference in Sedentary Behavior Minutes/Day
Description: difference between groups in minutes of sedentary behavior as captured by accelerometry
Time Frame: 12 months
Measure: Number; unit: adjusted minutes sedentary behavior/day
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 26 | 26
adjusted minutes sedentary behavior/day | 607 | 603

3. Secondary Outcome: Falls
Description: number of self-reported falls over 12 months/group
Time Frame: 12 months
Measure: Number; unit: number of falls over 12 months/group
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 27 | 26
number of falls over 12 months/group | 31 | 28

4. Secondary Outcome: Quality of Life (ICECAP-O)
Description: self-reported quality of life measure, scores range from 0 to 1 (0 = no capability, 1 = full capability); the higher the score the better.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 27 | 26
units on a scale | 0.81 (0.11) | 0.78 (0.13)

5. Secondary Outcome: Health Related Quality of Life (EQ5D-5L)
Description: self-reported health related quality of life (Visual Analogue Scale, 0 to 100). The higher the score means a better outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 27 | 26
units on a scale | 78.0 (15.5) | 77.2 (13.9)

6. Secondary Outcome: Lower Extremity Measure
Description: Self reported measure of lower extremity function. Scored 0 to 100. The higher the score the better.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 25 | 24
units on a scale | 82.27 (14.55) | 88.72 (9.40)

7. Secondary Outcome: Gait Speed (m/s)
Description: measurement of walking speed over 3 or 4 meters
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 27 | 26
m/s | 0.91 (0.47) | 0.90 (0.31)

8. Secondary Outcome: Grip Strength (Bilateral)
Description: measurement of grip strength using a dynamometer
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 25 | 23
kg | 25.64 (11.92) | 26.13 (10.25)

9. Secondary Outcome: Leg Strength (Fractured Leg)
Description: measurement of leg strength using a hand-held dynamometer
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 25 | 23
kg | 19.63 (7.55) | 18.87 (8.13)

10. Secondary Outcome: Timed up and Go (TUG)
Description: Measure of global mobility, reported in s. Participant is asked to rise from a chair, walk 3 meters, turn and walk back to chair and sit down.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 27 | 26
seconds | 16.1 (10.4) | 16.1 (9.5)

11. Secondary Outcome: Falls Self-efficacy International (FES-I)
Description: 16 items, the lower the score the better, e.g., more falls efficacy (range from 7-28)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 27 | 26
score on a scale | 12.1 (5.7) | 9.8 (3.1)

ADVERSE EVENTS:
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/26
Other Adverse Events (participants affected / at risk) | 0/27 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=27) | Intervention (N=26)
Possible adverse event (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — There was one serious adverse event (intervention group) that was possibly related to the intervention, but no follow-up action was required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No